CLINICAL TRIAL: NCT02070107
Title: A Phase 2 Clinical Trial of A Technology-Based Application To Improve The Triple Therapy Adherence Rate In Subjects With Chronic Genotype 1 Hepatitis C Infection
Brief Title: Technology-Based Application To Improve The Triple Therapy Adherence Rate In Subjects With Hepatitis C Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsored withdrew
Sponsor: University of Louisville (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Matthew Cave, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OICN130565
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no arms (Other): no arms, sponsor withdrew
  Interventions: Other: On Plan

INTERVENTIONS:
Other: On Plan — "On Plan" is a highly customizable software package developed by our co-investigator at the University of Louisville for a variety of applications related to compliance.

SUMMARY:
No more than 56% of subjects at the Robley Rex Louisville Veterans Administration Medical Center (VAMC) prescribed boceprevir-based triple therapy, will complete Hepatitis C (HCV) treatment as prescribed. Of patients who did not complete therapy, the primary reasons for discontinuation were side effects (48%) and non-adherence (32%). An intervention is needed to improve the treatment completion rate in subjects so they can achieve the high SVR rates noted in SPRINT-2 and RESPOND-2

DETAILED DESCRIPTION:
This protocol is a Phase II Open Label Clinical Trial of a technology-based application "On-Plan" (OP) which is expected to improve adherence to boceprevir-based triple therapy in subjects with chronic genotype 1 hepatitis C infection compared to historical controls from the University of Louisville. OP uses a combination of smart phone and computer-based social support to correct non-adherence and manage side effects as well as contingency management (positive reinforcement) when patient-reported compliance is documented by pill counts and/or electronic compliance monitors. 52 consenting subjects prescribed boceprevir-based triple therapy for chronic genotype 1 HCV according the U.S. prescribing information will be enrolled and all will receive the OP application. A Simon's two stage procedure will be utilized to minimize risk while preliminary efficacy/safety data are collected on this innovative "app" for HCV therapy.

ELIGIBILITY:
Inclusion Criteria:

The subject must meet ALL of the criteria listed below for entry:

1. Each subject must be willing and able to provide written informed consent for the trial.
2. Subjects must be willing to adhere to dose and visit schedules.
3. Each subject must be > 18years of age.
4. Each subject's weight must be ≥ 40 kg and ≤ 125 kg.
5. Subject must have previously documented HCV genotype 1 infection. Subjects with other or mixed genotypes are not eligible. The HCV-RNA result obtained from the central laboratory at the Screening Visit must confirm HCV genotype 1 infection with HCV RNA >10,000 IU/mL. Patients may be either treatment naïve or previously treated as long as they have not been treated with a protease inhibitor. Patients may have compensated cirrhosis.
6. Subject and subject's partner(s) must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study medication, or longer if dictated by local regulations. Postmenopausal women are not required to use contraception. Postmenopausal is defined as at least 12 consecutive months without a spontaneous menstrual period. Each sexually active male subject with a female partner(s) of child-bearing potential must also provide written informed consent to provide information regarding any pregnancy.

Exclusion Criteria:

The subject will be excluded from entry if ANY of the criteria listed below are met:

1. Subject is under the age of legal consent, is mentally or legally incapacitated, has significant emotional problems at the time of pre-study screening visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder which, in the opinion of the investigator, would interfere with the study procedures.
2. Subjects co-infected with the human immunodeficiency virus (HIV) or hepatitis B virus (Hepatitis B surface antigen [HBsAg] or HIV positive.
3. Treatment for hepatitis C with any investigational medication. Prior treatments with herbal remedies with known hepatotoxicity are exclusionary. All herbal remedies including but not limited to St. John's Wort (Hypericum perforatum) used for hepatitis C treatment must be discontinued before Day 1. Only silibinin based products such as silymarin (milk thistle) are allowed during the trial.
4. Subjects receiving any of the following medication(s) within 2 weeks prior to the Day 1 visit that are highly dependent on CYP3A4/5 for clearance, and for which elevated plasma concentrations could be associated with serious and/or life-threatening events such as orally administered midazolam, pimozide, amiodarone, flecainide, propafenone, quinidine, and ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine). The following medications are also exclusionary if taken within 2 weeks prior to the Day 1 visit: alfuzosin, cisapride, triazolam, sildenafil, and tadalafil (the latter 2 only if they are used for the indication of chronic obstructive pulmonary disease (COPD).
5. Participation in any other clinical trial within 30 days of the screening visit in this trial or intention to participate in another clinical trial during participation in this trial. Collection of additional blood, urine, or tissue samples or additional data, beyond that specified in this protocol, is prohibited (other than that related to the subject's medical care).
6. Evidence of decompensated liver disease.
7. Subject has evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC.
8. Subject is diabetic and/or hypertensive with clinically significant ocular examination findings within 6 months prior to the screening visit or between the screening visit and Day 1: retinopathy, cotton wool spots, optic nerve disorder, retinal hemorrhage, or any other clinically significant abnormality.
9. Subject has pre-existing psychiatric condition(s) including but not limited to: Current moderate or severe depression or history of severe psychiatric disturbance.
10. Subject has a clinical diagnosis of substance abuse which the investigators of the following specified drugs within specified timeframes:

    1. Alcohol, intravenous drugs, inhalational (not including marijuana), psychotropics, narcotics, cocaine use, prescription or over-the-counter drugs: within 1 year of the screening visit, OR
    2. Multi-drug abuse (e.g., two or more of the substances listed in Exclusion Criterion 10a within 3 years of screening visit, OR
    3. Subjects receiving opiate agonist substitution therapy within 1 year of screening visit (except for those subjects monitored in an opioid substitution maintenance program as specified in Section 7.3.5) OR
    4. Subject's historic marijuana use is deemed excessive by a physician investigator or is interfering with the subject's daily function. If subject's marijuana use is not deemed excessive and does not interfere with daily function, subject must be instructed to discontinue any current use of recreational marijuana prior to entry into trial and throughout the trial period.
11. Subject has any known medical condition that could interfere with the subject's participation in and completion of the trial, including, but not limited to:

    1. Central nervous system (CNS) trauma requiring intubation, intracranial pressure monitoring, brain meningeal or skull surgery, or resulting in seizure, coma, permanent neurologic deficits, abnormal brain imaging, or cerebral spinal fluid (CSF) leak. Prior brain hemorrhage and/or intracranial aneurysms (whether adequately repaired or not).
    2. Current uncontrolled seizure disorder unless now controlled on stable medical regimen that does not interact with boceprevir.
    3. History of stroke or transient ischemic attack.
    4. Immunologically mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], celiac disease, rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, sarcoidosis, severe psoriasis requiring oral or injected treatment, or symptomatic thyroid disorder).
    5. Clinically significant chronic pulmonary disease (e.g., clinical chronic obstructive pulmonary disease, interstitial lung disease, pulmonary fibrosis, sarcoidosis).
    6. Current or history of any clinically significant cardiac abnormalities/dysfunction (e.g., angina, congestive heart failure, myocardial infarction, pulmonary hypertension, complex congenital heart disease, cardiomyopathy, significant arrhythmia) including current uncontrolled hypertension, history of use of antianginal agents for cardiac conditions, or clinically significant abnormality on ECG performed at the pre-study screening visit.
    7. Any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial.
    8. Clinically significant gout within the last year.
    9. Clinically significant hemoglobinopathy, including, but not limited to, thalassemia major.
    10. Myelodysplastic syndromes.
    11. Coagulopathy, including, but not limited to, hemophilia.
    12. Organ transplants (including hematopoietic stem cell transplants) other than cornea and hair.
    13. Poor venous access that precludes routine peripheral blood sampling required for this trial.
    14. Subject with a history of gastric surgery (e.g., stapling, bypass) or subject with a history of malabsorption disorders (e.g., celiac sprue disease).

    p) Other serious medical condition which could be exacerbated by peg-IFN alfa-2a and/or RBV, in the opinion of the investigator.
12. Subject has evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin. Subjects under evaluation for malignancy are not eligible.
13. Female subject is pregnant, lactating, expecting to conceive or donate eggs OR Male subject is planning to impregnate or provide sperm donation or has a female sexual partner who is pregnant or is of childbearing potential and is unwilling to commit to using two methods of birth control throughout treatment and after the completion of all treatment (see Inclusion Criterion).
14. Subject has any other condition which, in the opinion of the principal investigator or physician, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study.
15. Subject had a life-threatening SAE during the screening period.
16. Subject is a member or a family member of the investigational study staff or sponsor staff directly involved with this study.

Laboratory Exclusion Criteria Note: If any of the laboratory exclusion criteria are met, the site may have the subject retested. If a single value is within 10% of the listed laboratory exclusion criterion value, and the value is considered not clinically significant by the investigator, the subject may be considered for enrollment. The value for platelets counts cannot be retested.

1. Hemoglobin <10 g/dL for females and <11 g/dL for males.
2. Neutrophils <1500/mm3, or <1,200/mm3 for subjects of African descent.
3. Platelets <60,000/mm3; this may not be retested and there is no variance allowed for this entry criteria.
4. Thyroid disorders:

   1. The subject may be enrolled if clinically euthyroid, AND
   2. The euthyroid function is confirmed by thyroxine/triiodothyronine (T4/T3) testing.
5. Serum glucose: Hemoglobin A1C >8.5%.
6. Positive pregnancy test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Treatment Completion | 24 weeks
  The percentage of patients completing treatment weeks 4, 8, 12, and 24 will be compared to historical controls treated with boceprevir-based triple therapy from our institution. In subjects not completing therapy as prescribed the reasons for discontinuation will be characterized including non-adherence and side effects and also compared to the historical controls.

SECONDARY OUTCOMES:
Virologic response | 24 weeks
  Virologic response to therapy will be determined at weeks 4, 8, 12, and 24; as well as at the end of treatment (EOTR) and 12 and 24 weeks after treatment completion (SVR12 and SVR24) and compared to historical controls. For these comparisons, subjects will be placed into appropriate subgroups (treatment naïve, relapsers, and non-responders). The percentage of subjects completing the entire course of therapy as initially prescribed will also be compared to historical controls. The percentage of subjects fulfilling the 80/80/80 rule will also be determined and their virologic outcomes determined although direct comparison with historical controls for these endpoints are our institution cannot be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cave, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States